CLINICAL TRIAL: NCT05370209
Title: A Prospective, Post-Market Clinical Follow-up Investigation to Verify Performance and Safety of Otinova® Ear Spray When Used in the Treatment of External Otitis Symptoms
Brief Title: Performance and Safety of Otinova® Ear Spray
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Circius Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIR_001
Record Dates: First submitted 2022-05-03; First posted 2022-05-11 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Otitis Externa
MeSH Terms: conditions — Otitis Externa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Otinova® Ear Spray (Experimental): Otinova® Ear Spray 1-2 sprays, twice daily for 7 days
  Interventions: Device: Otinova® Ear Spray

INTERVENTIONS:
Device: Otinova® Ear Spray — Ear spray

SUMMARY:
The purpose of this study is to assess the performance and safety of Otinova® Ear Spray when used in the treatment of external otitis symptoms.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will receive treatment with Otinova® Ear Spray for 7 days, twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 5 years old
* Clinical diagnosis of otitis externa based on otoscopic exam:

  a.Defined as a clinical score of at least 1, on a scale from 0 to 2 (none, mild/moderate, severe), for at least one of the OE signs (swelling, erythema and otorrhea)
* Ability to correctly administer Otinova as spray (not requiring tamponade), as judged by the Investigator
* Subject agrees to refrain from water immersion of the ears during the investigation
* Subject agrees to refrain from using other ear treatment products during the investigation
* For pediatric patients, provision of informed consent by subject and legal -Subject, and if applicable legal representative(s), are willing to comply with the protocol and attend all investigation visits.

Exclusion Criteria:

* Duration of OE signs/symptoms longer than 6 weeks
* Suspected perforated eardrum or eardrum fitted with drainage tube
* Post-mastoid surgery
* Prior otologic surgery within 6 months of enrollment (must be successfully healed)
* Conditions which may make it difficult to evaluate the therapeutic response (e.g malignant OE, abscess, granulation, polyps, congenital disorders)
* History of malignant tumors in the external ear canal, or currently receiving chemotherapy or radiation therapy
* Known allergy or sensitivity to any component of the device
* Use of topical or systemic antibiotics, corticosteroids or other treatment that could affect the study result within 7 days prior to enrolment
* Pregnancy or lactation at time of enrolment
* Subjects with any other condition that, as judged by the investigator, may make investigation procedures inappropriate
* Participation in another clinical investigation within 30 days of screening

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wilhelms, MD, PhD, Principal Investigator — Cordinator Medical Service AB; Sarah Ohlsson Maleki, MD, Principal Investigator — Öron-Näsa-Hals-Center Malmö
Locations (3):
- Sweden (3):
  - Carlanderska sjukhuset, Gothenburg
  - Cordinator Medical Service AB, Linköping
  - Öron-Näsa-Hals-Center Malmö, Malmo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Otinova® Ear Spray
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Otinova® Ear Spray
Number analyzed (Participants) | 28
Age, Customized [Count of Participants; unit: Participants]
  5-17 | 2
  >18 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 28

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure of Clinical Signs Swelling, Erythema and Otorrhea
Description: Proportion of subjects who have all signs of swelling, erythema and otorrhea scored as 0 on a scale from 0-2 (0=none, 1=mild/moderate, 2=severe) on Day 7
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Otinova® Ear Spray
Number analyzed (Participants) | 28
Participants | 28

2. Secondary Outcome: Change in Clinical Symptoms Itching, Otalgia and Tenderness
Description: Change in clinical symptoms itching, otalgia and tenderness, from Day 1 to Day 7, based on subject reported outcomes, using a score from 0 to 4, where 0 = no symptoms, 1= Mild, 2 = Moderate, 3= Severe and 4 = Very Severe
Time Frame: Change from Baseline (Day 1) to Day 7
Reporting Status: Not Posted

3. Secondary Outcome: Change in Microbes in the Earcanal
Description: Change of pathologic microbes in the ear canal from baseline (Day 1) to Day 7.
Time Frame: Change from Baseline (Day 1) to Day 7
Reporting Status: Not Posted

4. Secondary Outcome: Change of Moisture in the Earcanal
Description: Proportion of subjects who have signs of otorrhea (moisture) at baseline (Day 1)on a scale from 0-2 (0=none, 1=mild/moderate, 2=severe) and show an improvement of 1 or more points at Day 7.
Time Frame: Change from Baseline (Day 1) to Day 7
Reporting Status: Not Posted

5. Secondary Outcome: Change in Volume of Ear Canal
Description: Proportion of subjects who have signs of swelling at baseline (Day 1) on a scale from 0-2 (0=none, 1=mild/moderate, 2=severe) and show an improvement of 1 or more points at Day 7.
Time Frame: Change from Baseline (Day 1) to Day 7
Reporting Status: Not Posted

6. Secondary Outcome: User Handling
Description: Questionnaire regarding User handling - "How did you experience the use of the earspray?" and "Was it easy to apply the spray correctly in the ear?" using a 5-point scale: 1=very easy to use, 2=easy to use, 3=neither easy nor difficult to use, 4=difficult to use, 5=very difficult to use
Time Frame: Day 7
Reporting Status: Not Posted

7. Secondary Outcome: Change in Sleep
Description: Proportion of subjects with less sleep disruption Day 7 compared to baseline (Day 1), as reported in subject diary
Time Frame: Change from Baseline (Day 1) to Day 7
Reporting Status: Not Posted

8. Secondary Outcome: Chnage in Pain Relief Medication Use
Description: Proportion of subjects with less use of pain relief medication for ear pain on Day 7 compared to baseline (Day 1), as reported in subject diary
Time Frame: Change from Baseline (Day 1) to Day 7
Reporting Status: Not Posted

9. Secondary Outcome: Antibiotic Use
Description: Use of antibiotics for OE symptoms at Day 7
Time Frame: Day 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | Otinova® Ear Spray
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otinova® Ear Spray (N=28)
Pain in ear (Ear and labyrinth disorders) | 2 (2)
Pain in arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomach flu (Gastrointestinal disorders) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to slow recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT05370209/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT05370209/SAP_001.pdf